CLINICAL TRIAL: NCT04148092
Title: Expanded Access Program for Ripretinib in Patients With Locally Advanced Unresectable or Metastatic GIST Who Have Received Treatment With Prior Therapies
Brief Title: Expanded Access Program of Ripretinib (DCC-2618) for the Treatment of Patients With Advanced GIST
Status: Approved for marketing | Type: Expanded Access
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DCC-2618-99-001
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: GIST - Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: ripretinib — orally administered solid dosage form
  Other Names: DCC-2618

SUMMARY:
This is an open-label, single-arm, multicenter expanded access study to provide patients who have locally advanced unresectable or metastatic gastrointestinal stromal tumor (GIST) and have received treatment with at least 2 prior Food and Drug Administration (FDA)-approved therapies early access to ripretinib until such time that ripretinib becomes commercially available or the Sponsor chooses to discontinue the program.

DETAILED DESCRIPTION:
The EAP is no longer enrolling patients in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ≥ 18 years of age at the time of informed consent
2. Histologic diagnosis of GIST
3. Patients must have received prior treatment with at least 2 of the FDA-approved drugs for GIST: imatinib, sunitinib, and regorafenib.
4. Female patients of childbearing potential must have a negative pregnancy test at Screening.
5. Patients of reproductive potential must agree to follow the contraception requirements.
6. Patient is capable of understanding and complying with the protocol and has signed the ICF. A signed ICF must be obtained before any study specific procedures are performed.
7. Adequate organ function and bone marrow reserve as determined by the Investigator at Screening.
8. Resolution to Grade 1 or baseline of all serious toxicities from prior therapy prior to initiating treatment with ripretinib

Exclusion Criteria:

1. Eligible to participate in another ongoing clinical study in which the patient may have access to ripretinib
2. Received treatment with anticancer therapy, including investigational therapy, or investigational procedures within 7 days or 5 × the half-life (whichever is longer) prior to the first dose of ripretinib. For prior biological therapies (eg, monoclonal antibodies with a half-life longer than 3 days), the interval must be at least 28 days prior to the first dose of ripretinib.
3. Received prior treatment with ripretinib
4. Known active central nervous system metastases
5. With a concurrent malignancy for which treatment is being received that may interfere with the potential benefits of ripretinib to the patient
6. Undergone major surgeries (eg, abdominal laparotomy) within 4 weeks of the first dose of ripretinib. Following major surgeries, > 4 weeks prior to the first dose of ripretinib, all surgical wounds must be healed and free of infection or dehiscence.
7. Any other clinically significant comorbidities which in the judgment of the Investigator, could predispose the patient to safety risks
8. Known human immunodeficiency virus or hepatitis C infection only if the patient is taking medications that must be avoided or taken with caution per protocol, active hepatitis B, or active hepatitis C infection
9. If female, the patient is pregnant or lactating.
10. Known allergy or hypersensitivity to any component of the investigational product. Patients with a history of Stevens-Johnson syndrome on a prior tyrosine kinase inhibitor are excluded.
11. Gastrointestinal abnormalities including but not limited to:

    * inability to take oral medication
    * malabsorption syndromes
    * requirement for intravenous alimentation
12. Any active bleeding excluding hemorrhoidal or gum bleeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- See also: Ripretinib EAP Webpage — https://www.deciphera.com/pipeline/expanded-access/